CLINICAL TRIAL: NCT02290834
Title: Chemotherapy-induced Cognitive and Brain Changes in Older Adults With Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Michael W Parsons, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-217
Record Dates: First submitted 2014-11-05; First posted 2014-11-14 (Estimated); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Impaired Cognition; Chemo-brain; Breast Cancer
Keywords: Chemotherapy related cognitive impairment; Chemo-brain
MeSH Terms: conditions — Cognition Disorders; Breast Neoplasms; Chemotherapy-Related Cognitive Impairment | interventions — Functional Status; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ARM 1 (Active Comparator): Breast cancer patients treated with chemotherapy
  * Cognitive, functional and subjective assessments (Pre and Post Treatment)
  * Imaging (Pre and Post Treatment)
    * Magnetic Resonance Imaging (MRI) Scan
    * Magnetic Resonance Imaging (MRI) Scan / Positron Emission Tomography (PET) Scan
  Interventions: Other: Cognitive, functional and subjective assessments; Device: MRI; Radiation: PET Scan
- ARM 2 (Active Comparator): Non-treated breast cancer patient control
  * Cognitive, functional and subjective assessments (Post enrollment and 6-14 months later
  * Imaging (Post Enrollment and at 8-14 months later)
    * Magnetic Resonance Imaging (MRI) Scan
    * Magnetic Resonance Imaging (MRI) Scan / Positron Emission Tomography (PET) Scan
  Interventions: Other: Cognitive, functional and subjective assessments; Device: MRI; Radiation: PET Scan
- ARM 3 (Active Comparator): Healthy control subjects
  * Cognitive, functional and subjective assessments (Post enrollment and 6-14 months later
  * Imaging (Post Enrollment and at 8-14 months later)
    * Magnetic Resonance Imaging (MRI) Scan
    * Magnetic Resonance Imaging (MRI) Scan / Positron Emission Tomography (PET) Scan
  Interventions: Other: Cognitive, functional and subjective assessments; Device: MRI; Radiation: PET Scan

INTERVENTIONS:
Other: Cognitive, functional and subjective assessments — Cognitive and functional assessments
Device: MRI — Magnetic Resonance Imaging (MRI) Scan
Radiation: PET Scan — Positron Emission Tomography (PET) Scan

SUMMARY:
This research study evaluates the effect of chemotherapy on cognition (thinking) and the brain in people with breast cancer.

DETAILED DESCRIPTION:
* This study is being done to study effects of chemotherapy (cancer treatment) on the brain and cognition (thinking). "Chemo-brain" is a term sometimes used to refer to effects of chemotherapy on the brain and cognition (thinking).
* This study is being done to test for "chemo-brain" in older adults with breast cancer treated with chemotherapy, and to identify people who are most likely to be affected. The investigators will look at thinking abilities and brain images before and after chemotherapy to see if it can help identify people at risk for cognitive side effects of the treatment, and to better understand effects of treatment on brain structure and function.
* The investigators are looking for participants who have either been recently recently diagnosed breast cancer participant or a healthy volunteer.
* What is involved in the study:

  * Memory and Thinking Tests
  * Imaging: Either MRI/or MRI and PET Scans

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients treated with chemotherapy- Group 1 (experimental group)

  * Participants must meet the following criteria on screening examination to be eligible to participate in the behavioral +/- imaging components of study
  * New diagnosis histologically confirmed invasive breast cancer
  * Treatment plan to include chemotherapy
  * Female subjects age ≥ 60 years.
  * Life expectancy ≥ 1 year
  * Karnofsky Performance Score (KPS) ≥ 80
  * Ability to understand and the willingness to sign a written informed consent document.
* Non-treated breast cancer patient controls- Group 2 (control group)

  * Participants must meet the following criteria on screening examination to be eligible to participate in the behavioral +/- imaging components of study:
  * New diagnosis histologically confirmed invasive breast cancer
  * Treatment plan does not include chemotherapy
  * Age ≥ 60 years.
  * Life expectancy ≥ 1 year
  * Karnofsky Performance Score (KPS) ≥ 80
  * Ability to understand and the willingness to sign a written informed consent document.
* Healthy control subjects- Group 3 (control group)

  * Participants must meet the following criteria on screening examination to be eligible to participate in the behavioral +/- imaging components of study:
  * Age ≥ 60 years.
  * Life expectancy ≥ 1 year
  * Karnofsky Performance Score (KPS) ≥ 80
  * Ability to understand and the willingness to sign a written informed consent document.
  * Participants with well-controlled vascular risk factors, such as treated hypertension, treated hyperlipidemia or well-controlled Type II diabetes (glucose levels <250) may be included.
  * Serum Pregnancy Testing: STAT quantitative serum hCG pregnancy testing for all women of childbearing potential. Imaging will not start until and unless the test result returns negative.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study:

  * Participants with clinical or radiographic evidence of metastatic CNS disease
  * Subjects with MMSE scores below 24
  * Active or history of major psychiatric disorders such as schizophrenia, schizoaffective disorder, major affective disorder in mid-life, or treatment with ECT (Mild depression that is well treated with stable dose of SSRI antidepressants may be allowed).
  * Substance abuse within the past 2 years
  * Huntington's disease, hydrocephalus or seizure disorder
* In addition to exclusion criteria above, participants who exhibit any of the following conditions at screening will not be eligible for admission into imaging portion of the study:

  * Participants with contraindications to MRI (i.e., implanted metal including pacemakers, cerebral spinal fluid shunts, aneurysm clips, artificial heart valves, ear implants or metal/foreign objects in the eyes and those with a history of claustrophobia), injuries to the eyes with metal without X-ray documentation that metal was removed

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-03; Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive performance scores | Baseline, immediately after completion of chemo, and 6 months after completion of chemotherapy

SECONDARY OUTCOMES:
Correlation between baseline amyloid accumulation in the brain and change in cognitive performance | Baseline, 6 months after completion of chemotherapy
Correlation between baseline tau accumulation in the brain and change in cognitive performance | Baseline, 6 months after completion of chemotherapy
Correlation between change in tau accumulation in the brain (from baseline to 6 months after completion of chemotherapy) and change in cognitive performance (from baseline to 6 months after completion of chemotherapy) | Baseline, 6 months after completion of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Michael Parsons, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Massachusetts General Hospital/North Shore Cancer Center, Salem, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided
No data are yet available